CLINICAL TRIAL: NCT01553695
Title: Validation of a Clinical Interview for a Diagnosis of ADHD in Adults. Cross-validity of Screening Instruments ADHD in Adults. Estimation of Prevalence in France
Brief Title: Adults With Attention Deficit Hyperactivity Disorder (ADHD): Validation of a Clinical Interview and Screening Instruments in French
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 11-AOI-01
Record Dates: First submitted 2012-01-26; First posted 2012-03-14 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2012-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Touble; deficit; attention; hyperactivity; Touble deficit attention with hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- general population (Active Comparator)
  Interventions: Other: questionary
- ADHD Patient (Experimental)
  Interventions: Other: questionary

INTERVENTIONS:
Other: questionary — Subjects have to fill out a booklet of questionnaires
  Arms: general population
Other: questionary — Subjects have to fill out a booklet of questionnaires
  Arms: ADHD Patient

SUMMARY:
ADHD is a neurodevelopmental disorder that affects about 5% of school-age children and 3.5% of adults worldwide. This condition is under-recognised in France and other European countries and, therefore, under-diagnosed.

As part of the European Network for Adult ADHD, the investigators translated into French a structure interview called the Diagnostic Interview for Adult ADHD (DIVA). The investigators also translated rating scales such as the ASRS and the WURS. Validation studies are rare in France.

The aim of this study is to include two groups of 50 adults whether they have or not ADHD with respect of Diagnostic and Statistical Manual - Revision 4(DSM-IV) criteria as implemented in the DIVA (i.e. actual at adulthood and past in childhood). Subjects have to fill out a booklet of questionnaires including the WHO's Adult ADHD Symptom Rating Scale (ASRS) (screening tool for actual diagnosis) and the Wender Utah Rating Scale (WURS, a screening tool for ADHD in childhood with respect of the Utah criteria). The investigator will be able to compare the actual criteria for ADHD between the ASRS and the DIVA, and the past criteria for ADHD between the WURS and the DIVA. Finally, an estimate of the prevalence of ADHD in adults will be computed.

ELIGIBILITY:
Inclusion Criteria:

* Authorization to use the data signed social security affiliation

Exclusion Criteria:

* Patient presenting a known neurological or psychiatric disorder, or a deficit Intellectual because the attentional disorders(confusions), the psychomotor excitement and The impulsiveness can be symptoms inherent to the other pathologies Neurological and\or psychiatric.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic of ADHD using DSM-IV criteria as implemented in the DIVA | Baseline

SECONDARY OUTCOMES:
score of rating scales (ASRS and WURS) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Herve CACI, PH, Principal Investigator — CHU de Nice- GCS Lenval
Locations (1):
- Pediatric Hospital Lenval, Nice, France